CLINICAL TRIAL: NCT01566357
Title: Impact of Milk and Casein Phosphopeptide-amorphous Calcium Phosphate on Erosion/Abrasion of Enamel and Dentin - an in Situ Study
Brief Title: Impact of Milk on Erosion/Abrasion of Enamel and Dentin - an in Situ Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Borrow Foundation (Unknown)
Responsible Party: Principal Investigator, Annette Wiegand, PD Dr. med. dent., PD Dr. med. dent., University of Zurich
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 029/UZS
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Erosion Protection
Keywords: dental erosion; enamel; dentin
MeSH Terms: conditions — Tooth Erosion | interventions — Toothpastes; Milk; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Fluoride-free toothpaste (No Intervention)
- Fluoride toothpaste (Active Comparator)
  Interventions: Other: Toothpaste
- Milk (Active Comparator)
  Interventions: Dietary Supplement: Milk
- Fluoridated milk (Active Comparator)
  Interventions: Dietary Supplement: Fluoridated Milk
- CPP-ACP (Active Comparator)
  Interventions: Drug: Tooth Mousse
- Fluoridated CPP-ACP (Active Comparator)
  Interventions: Drug: MI Paste Plus
- Fluoride mouthrinse (Active Comparator)
  Interventions: Drug: Elmex Erosion Protection

INTERVENTIONS:
Other: Toothpaste
  Arms: Fluoride toothpaste
Dietary Supplement: Milk
  Arms: Milk
Dietary Supplement: Fluoridated Milk
  Arms: Fluoridated milk
Drug: Tooth Mousse
  Arms: CPP-ACP
Drug: MI Paste Plus
  Arms: Fluoridated CPP-ACP
Drug: Elmex Erosion Protection
  Arms: Fluoride mouthrinse

SUMMARY:
This in situ study aims to investigate

* the protective potential of milk and fluoridated milk on erosive wear of enamel
* the protective potential of milk and fluoridated milk on erosive wear of dentin
* to compare to protective potential of milk and fluoridated milk with products containing casein phosphopeptide-amorphous calcium phosphate
* to compare the protective potential of milk and fluoridated milk with a fluoridated toothpaste or stannous-chloride containing fluoride solution (SnCl2/AmF/NaF)

DETAILED DESCRIPTION:
Dental erosion is defined as the pathogenic, chronic, chemical removal of dental hard tissues due to the frequent contact to extrinsic or intrinsic acids. The dissolution process is determined by the pH, the chelating properties, mineral content and kind of acid, but in the same time modified by various biological (e.g. saliva, pellicle) and behavioural factors.

The anticariogenic properties of milk are widely investigated, but information of the effects of milk or milk components on the development of erosion are limited. It is suggested that the demineralisation process is reduced by the presence of calcium and phosphate, but also that casein proteins affect the demineralisation by adsorbing to the hydroxyapatite surface and inhibiting its dissolution. Initial studies suggest that milk is able to increase rehardening of acid-softened enamel, but information about the effects of milk on dentin erosion are not available yet. Particularly, the effect of fluoridated milk on dental erosion was not investigated yet.

In contrast, recent studies analysed the effects of products containing casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) on erosion, as it is suggested that CPP-ACP promotes a supersaturated state and increased remineralisation of demineralised dental hard tissue. However, in situ studies on the effect of CPP-ACP on erosion are limited to one study, which compared microhardness of enamel after treatment with CPP-ACP and CPP-ACP and 900 ppm fluoride, but failed to use appropriate controls in form of other products containing calcium and phosphate or fluoride. In summary, the effects of milk, in particular fluoridated milk, and products containing milk proteins, such as casein phosphopeptide-amorphous calcium phosphate, on erosive wear were not analysed in an in-situ-model so far.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* non-treated caries lesions
* orthodontic treatment which does not allow to wear an intraoral device
* hyposalivation
* allergy against milk or milk proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Substance loss (profilometry) | after each study phase (5 days)
  Each intervention will be tested for 5 days in situ. Then, enamel or dentin loss, respectively, will be determined by profilometry

CONTACTS AND LOCATIONS:
Overall Officials: Annette Wiegand, PD Dr. med. dent., Principal Investigator — University of Zurich, Switzerland; Thomas Attin, Prof. Dr. med. dent., Study Director — University of Zurich, Switzerland
Locations (1):
- Clinic for Preventive Dentistry, Periodontology and Cariology, University of Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Wiegand A, Muller I, Schnapp JD, Werner C, Attin T. Impact of fluoride, milk and water rinsing on surface rehardening of acid softened enamel. An in situ study. Am J Dent. 2008 Apr;21(2):113-8. PMID 18578180
- [Background] Hemingway CA, White AJ, Shellis RP, Addy M, Parker DM, Barbour ME. Enamel erosion in dietary acids: inhibition by food proteins in vitro. Caries Res. 2010;44(6):525-30. doi: 10.1159/000320984. Epub 2010 Oct 28. PMID 20980757
- [Background] White AJ, Gracia LH, Barbour ME. Inhibition of dental erosion by casein and casein-derived proteins. Caries Res. 2011;45(1):13-20. doi: 10.1159/000322300. Epub 2010 Dec 11. PMID 21160185
- [Background] Wiegand A, Hiestand B, Sener B, Magalhaes AC, Roos M, Attin T. Effect of TiF4, ZrF4, HfF4 and AmF on erosion and erosion/abrasion of enamel and dentin in situ. Arch Oral Biol. 2010 Mar;55(3):223-8. doi: 10.1016/j.archoralbio.2009.11.007. Epub 2010 Jan 18. PMID 20083245
- [Derived] Wiegand A, Attin T. Randomised in situ trial on the effect of milk and CPP-ACP on dental erosion. J Dent. 2014 Sep;42(9):1210-5. doi: 10.1016/j.jdent.2014.07.009. Epub 2014 Jul 17. PMID 25038509